CLINICAL TRIAL: NCT00001237
Title: Pilot Protocol for the Treatment of Patients With Small Non-Cleaved and Diffuse Large Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 890041; 89-C-0041
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Burkitt Lymphoma; Lymphoma, Large-Cell, Diffuse; Lymphoma, Small Noncleaved-Cell
Keywords: Burkitt's Lymphoma; GM-CSF; High-Grade
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: granulocyte-macrophage colony stimulating factor (GM-CSF)

SUMMARY:
Major improvements in the treatment of childhood non-lymphoblastic lymphomas have taken place in the last ten years. Though the survival rate in low risk patients (i.e., those with stage I & II disease and serum LDH of less than 350 IU/dL) was as high as 90% with the previous Pediatric Branch protocol, only 32% of patients in the high risk group achieved long term remission. The present protocol is designed to improve survival in the high risk group by using alternating non-cross resistant drug regimens. We plan to determine whether using granulocyte-macrophage colony stimulating factor (GM-CSF) in this group would increase dose-intensity and ameliorate myelotoxicity. We also plan to study the effect on survival of decreasing the duration of treatment to three months from the present year-long therapy in low-risk patients.

DETAILED DESCRIPTION:
Major improvements in the treatment of childhood non-lymphoblastic lymphomas have taken place in the last ten years. Though the survival rate in low risk patients (i.e., those with stage I & II disease and serum LDH of less than 350 IU/dL) was as high as 90% with the previous Pediatric Branch protocol, only 32% of patients in the high risk group achieved long term remission. The present protocol is designed to improve survival in the high risk group by using alternating non-cross resistant drug regimens. We plan to determine whether using granulocyte-macrophage colony stimulating factor (GM-CSF) in this group would increase dose-intensity and ameliorate myelotoxicity. We also plan to study the effect on survival of decreasing the duration of treatment to three months from the present year-long therapy in low-risk patients.

ELIGIBILITY:
High Risk Protocol: Patients with small non-cleaved (Burkitt or Burkitt-like) or diffuse large cell lymphomas except those with:

a) Minimal extra-abdominal tumor as the sole site of disease and a serum LDH less than 1.5 times the upper limit of normal (NIH patients, less than 350 U/L) or except those with b) completely resected small, localized abdominal mass (involved segmental lymph nodes permitted) and a serum LDH level less than 1.5 times upper limit of normal (NIH patients less than 350 U/L).

All patients with small non-cleaved (Burkitt or Burkitt-like) or diffuse large cell lymphomas with a serum LDH level greater than 1.5 times the upper limit of normal (NIH patients, greater than 350 U/L), regardless of the clinically documented extent of disease.

All patients with small non-cleaved (Burkitt or Burkitt-like) or diffuse large cell lymphomas with testicular involvement.

Low risk protocol: Patients with small non-cleaved (Burkitt or Burkitt-like) or diffuse large cell lymphomas with a) minimal extra-abdominal disease as the sole site of disease and a serum LDH less than 1.5 times the upper limit of normal (NIH patients, less than 350 U/L) or b) completely resected small, localized abdominal mass (involved segmental lymph nodes permitted for gastrointestinal disease) and a serum LDH level less than 1.5 times the upper limit of normal (NIH patients, less than 350 U/L).

No patients with lymphoblastic lymphomas, low grade or follicular lymphomas.

No patients with peripheral T cell lymphomas that do not fall into the category of anaplastic large cell lymphoma.

No patients with a previously documented lymphoma or histological evidence of co-existing lymphoma of other histology.

No patients who have been previously treated with chemotherapy or radiotherapy.

No patients with HIV infection.

No patients above the age of 60 years.

No patients with a history of inherited or non-HIV acquired immunodeficiency syndromes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1989-03; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Magrath I, Barriga F, McManaway M, Shiramizu B. The molecular analysis of chromosomal translocations as a diagnostic, epidemiological and potentially prognostic tool in lymphoid neoplasia. J Virol Methods. 1988 Sep;21(1-4):275-89. doi: 10.1016/0166-0934(88)90073-0. PMID 3053744
- [Background] Pelicci PG, Knowles DM 2nd, Magrath I, Dalla-Favera R. Chromosomal breakpoints and structural alterations of the c-myc locus differ in endemic and sporadic forms of Burkitt lymphoma. Proc Natl Acad Sci U S A. 1986 May;83(9):2984-8. doi: 10.1073/pnas.83.9.2984. PMID 3458257
- [Background] Magrath IT, Janus C, Edwards BK, Spiegel R, Jaffe ES, Berard CW, Miliauskas J, Morris K, Barnwell R. An effective therapy for both undifferentiated (including Burkitt's) lymphomas and lymphoblastic lymphomas in children and young adults. Blood. 1984 May;63(5):1102-11. PMID 6546890